CLINICAL TRIAL: NCT01030809
Title: A Cluster Randomized Controlled Trial of a Treatment Algorithm for the Management of Crohn's Disease
Brief Title: Trial of a Treatment Algorithm for the Management of Crohn's Disease
Acronym: REACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP0901
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; community based gastroenterology practices Canada and Belgium; Cluster randomization controlled trial; Remission; Corticosteroids; Documented diagnosis of Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care practice (No Intervention): Patients managed according to usual care practices
- Treatment Algorithm (Active Comparator): Practitioners assigned to the intervention arm will be educated on the use of the treatment algorithm.
  Interventions: Other: Treatment Algorithm for Crohn's Disease

INTERVENTIONS:
Other: Treatment Algorithm for Crohn's Disease — Practitioners assigned to the intervention arm will be educated on the use of the treatment algorithm.
  Arms: Treatment Algorithm

SUMMARY:
Assess if the implementation of a treatment algorithm will improve the management of Crohn's disease (CD) in comparison to usual care based gastroenterology practices.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic inflammatory disorder of the gastrointestinal tract. During disease exacerbations, pharmacological or surgical intervention is usually needed to re-establish remission. Ideally, strategies should be employed to maintain patients in long-term remission while minimizing exposure to corticosteroids and reduce therapy-related toxicity.

Nevertheless, in reality many patients with CD do not receive effective therapy and their disease often remains active, leading to uncontrolled inflammation and complications from either the underlying disease or corticosteroids. Although treatment guidelines exist, they do not adequately define treatment goals and the duration of treatment cycles is not specified Optimizing outcomes in CD requires rapid control of inflammation. Intuitively, persistent inflammation leads to persistent symptoms, tissue damage, and disease-related complications. Conventional therapy is frequently ineffective in moderate to severe CD, and is often continued for a prolonged time. Consequently, many patients are under-treated. An alternate strategy that minimizes the use of corticosteroids and encourages the earlier use of immunosuppressive agents and tumour necrosis factor (TNF) antagonists may be optimal. However it is unknown whether this approach is superior to usual care

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Crohn's disease
* Able to speak and understand English, French or Flemish
* Access to a telephone or email/internet service
* Written informed consent must be obtained and documented

Exclusion Criteria:

* Any conditions (e.g., history of alcohol or substance abuse) which in the opinion of the investigator , may interfere with the patients ability to comply with study procedures
* Participating in other investigational studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1999 (Actual)
Dates: Start 2010-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in remission at the end of the 24 month followup period. Remission is defined as a HBS< or = 4 without use of steroids for the treatment of CD. the primary analysis will be performed at the level of the practice. | 24 months

SECONDARY OUTCOMES:
Proportion of patients in remission over study, change in mean HBS; use of CD meds, occurrence of surgery/hospitalization for CD and complications, patients' health related QOL measured by SF-36 & EQ-5D; physician/patient satisfaction with therapy. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Feagan, MD, Principal Investigator — Robarts Research Institute - University of Western Ontario
Locations (1):
- Robarts Clinical Trials, Robarts Research Institute, London, Ontario, Canada

REFERENCES:
- [Derived] Singh S, Stitt LW, Zou G, Khanna R, Dulai PS, Sandborn WJ, Feagan BG, Jairath V. Early combined immunosuppression may be effective and safe in older patients with Crohn's disease: post hoc analysis of REACT. Aliment Pharmacol Ther. 2019 May;49(9):1188-1194. doi: 10.1111/apt.15214. Epub 2019 Mar 19. PMID 30891808
- [Derived] Khanna R, Bressler B, Levesque BG, Zou G, Stitt LW, Greenberg GR, Panaccione R, Bitton A, Pare P, Vermeire S, D'Haens G, MacIntosh D, Sandborn WJ, Donner A, Vandervoort MK, Morris JC, Feagan BG; REACT Study Investigators. Early combined immunosuppression for the management of Crohn's disease (REACT): a cluster randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1825-34. doi: 10.1016/S0140-6736(15)00068-9. Epub 2015 Sep 3. PMID 26342731